CLINICAL TRIAL: NCT05704621
Title: A Randomized Phase II Study of Secondary Cytoreductive Surgery (CRS) in Patients With Relapsed Ovarian Cancer Who Have Progressed on PARP Inhibitor Maintenance
Brief Title: Secondary Cytoreductive Surgery (CRS) in Patients With Relapsed Ovarian Cancer Who Have Progressed on PARP Inhibitor Maintenance
Acronym: SOCCER-P
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Korea University Guro Hospital (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry); Chong Kun Dang Pharmaceutical Corp. (Industry); Yonsei University (Other); KGOG: Korean Gynaelogical Onology Group, Korea (Unknown); Japanese Gynecologic Oncology Group (Other); Asia-Pacific Gynecologic Oncology Trials Group (APGOT) (Unknown)
Responsible Party: Principal Investigator, Hyun Woong Cho, Assistant professor, Korea University Guro Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KGOG3067/JGOG3036/APGOT-OV11
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Ovarian Cancer; Drug Related Neoplasm/Cancer
Keywords: recurrent ovarian cancer; PARP inhibitor resistance; secondary cytoreductive surgery; progression during PARP inhibitor maintenance
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: A randomized superiority trial (Surgery versus No Surgery)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- secondary cytoreductive surgery followed by chemotherapy (Experimental): surgery arm
  Interventions: Procedure: secondary cytoreductive surgery; Drug: chemotherapy
- chemotherapy (Active Comparator): no surgery arm
  Interventions: Drug: chemotherapy

INTERVENTIONS:
Procedure: secondary cytoreductive surgery — Maximum effort cytoreductive surgery
  Other Names: secondary cytoreductive surgery followed by chemotherapy
  Arms: secondary cytoreductive surgery followed by chemotherapy
Drug: chemotherapy — six cycles of platinum-based chemotherapy +/- bevacizumab
  Other Names: no surgery and only chemotherapy

SUMMARY:
This is a randomized phase II study of secondary cytoreductive surgery (CRS) in patients with relapsed ovarian cancer who have progressed on PARP inhibitor maintenance.

DETAILED DESCRIPTION:
The primary objective is to find out whether the CRS is beneficial in patients who have progressed on PARPi maintenance.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first recurrence of platinum sensitive, invasive epithelial ovarian-, fallopian tube- or primary peritoneal cancer of any initial stage.
* Progression-free interval of at least 6 months after end of last platinum- containing therapy,
* Progressed during PARP inhibitor maintenance
* Women aged ≥ 18 years
* Complete resection of the tumor seems possible (estimated by an experienced surgeon). Intra-abdominal disease has to be excluded by MRI/CT, if other surgical approaches for isolated extra-abdominal recurrences are planned

  1. A positive AGO-score or iMODEL+PET/CT
  2. Patients who are likely to be completely resected according to the investigator's judgment will be allowed by consensus between PI(surgeon) and designated radiologist even if AGO or iMODEL+PET/CT negative.
* Patients who have given their signed and written informed consent and their consent to data transmission and -processing.

Exclusion Criteria:

* Patients with non-epithelial tumors as well as borderline tumors.
* Patients without recurrence who are scheduled for diagnostic/second-look surgery or debulking surgery after completion of chemotherapy
* More than one prior chemotherapy
* Patients with second, third, or later recurrence
* Patients with second malignancies who have been treated by laparotomy, as well as other neoplasms, if the treatment might interfere with the treatment of relapsed ovarian cancer or if major impact on prognosis is expected.
* Patients with so-called platinum-refractory tumor, i.e. progression during chemotherapy or recurrence within 6 months after end of former first platinum- containing therapy
* Only palliative surgery planned
* Radiological signs suggesting metastases not accessible to surgical removal (i.e. complete resection is deemed impossible)
* Any concomitant disease not allowing surgery and/or chemotherapy
* Any medical history indicating excessive peri-operative risk
* Any current medication inducing considerable surgical risk (e.g. bleeding: due to oral anticoagulating agents, bevacizumab)
* No assessable archival tumor tissue

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-28 (Estimated); Study Completion 2028-12-28 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | Up to 2 year
  interval between date of randomization and the date of second relapse/progression or death, whatever occurs first

SECONDARY OUTCOMES:
Overall survival | Up to 2 year
  from date of randomisation until death

OTHER OUTCOMES:
30-day post-operative complications | From the operation until after 30 days
  MSKCC surgical complications grading method and CTCAE v4.03 criteria will be adopted for evaluating the perioperative complications
Time to first subsequent anticancer therapy | Up to 1 year
  From date of randomization until the date of first recurrent anticancer therapy
Time to second subsequent anticancer therapy | Up to 2 year
  From date of randomization until the date of secondary recurrent anticancer therapy
Quality of life | baseline, 6 month and 1year after randomization
  EORTC QLQ-C30,OV28, and EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Hyun-Woong Cho, MD. PhD., Principal Investigator — Korea University Guro Hospital
Locations (1):
- Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho HW, Kim HS, Park JY, Lee YY, Lim MC, Lee SJ, Min KJ, Eoh KJ, Lee KB, Kim MK, Song JY, Shim SH, Ji YI, Song YJ, Chang SJ, Kim MK, Abe A, Kobayashi Y, Kajiyama H, Shimada M, Okamoto A, Ng JS, Lee JY. A randomized phase II study of secondary cytoreductive surgery in patients with relapsed ovarian cancer who have progressed on a PARP inhibitor as first-line maintenance therapy: the SOCCER-P study (KGOG 3067/JGOG 3036/APGOT-OV11). Int J Gynecol Cancer. 2024 Nov 4;34(11):1809-1812. doi: 10.1136/ijgc-2024-005838. PMID 39164041